CLINICAL TRIAL: NCT07229092
Title: Comparison of Serratus Plane Block and Rhomboid Intercostal Plane Block for Postoperative Analgesia in Patients Undergoing Breast Reduction Surgery: A Randomized Clinical Study
Brief Title: Comparison of Serratus Plane Block and Rhomboid Intercostal Plane Block for Postoperative Analgesia in Breast Reduction Surgery
Acronym: SAPB-RIPB
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Konul Karaja (Other)
Responsible Party: Sponsor-Investigator, Konul Karaja, Anesthesiology Research Fellow / MD, Aydin Adnan Menderes University
Organization: Aydin Adnan Menderes University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ADU-SAPB-RIPB-2025
Record Dates: First submitted 2025-11-13; First posted 2025-11-14 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Postoperative Analgesia in Breast Reduction Surgery; Postoperative Pain; Postoperative Pain Breast Reduction; Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: The study includes two parallel groups. Patients undergoing breast reduction surgery will be randomly assigned to receive either ultrasound-guided serratus plane block (SPB) or rhomboid intercostal plane block (RIPB) for postoperative analgesia.
Who Masked: Participant, Outcomes Assessor
Masking Description: The patients and the outcome assessor who recorded postoperative pain scores were blinded to the type of block performed
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Serratus Plane Block (Experimental): "Patients in this group will receive an ultrasound-guided serratus anterior plane block (SAPB) before induction of general anesthesia, while awake. A total of 30 mL of local anesthetic solution (5 mL normal saline, 5 mL of 2% lidocaine, and 20 mL of 0.25% bupivacaine) will be prepared. The total solution will be divided equally between both breasts, with 15 mL administered to the right side and 15 mL to the left side. Each side will receive a single injection point along the midaxillary line to provide adequate spread within the serratus plane.
  Interventions: Procedure: Serratus Plane Block
- Rhomboid Intercostal Plane Block (Active Comparator): "Patients in this group will receive an ultrasound-guided rhomboid intercostal plane block (RIPB) before induction of general anesthesia, while awake. A total of 30 mL of local anesthetic solution (5 mL normal saline, 5 mL of 2% lidocaine, and 20 mL of 0.25% bupivacaine) will be prepared. The total solution will be divided equally between both breasts, with 15 mL administered on the right and 15 mL on the left. Each side will receive a single injection point beneath the medial border of the scapula at the level of the intercostal plane to ensure adequate spread between the rhomboid major muscle and intercostal muscles."
  Interventions: Procedure: Rhomboid Intercostal Plane Block (RIPB)
- Control Group (No Block) (Other): Patients in this group will not receive any regional block. Standard general anesthesia and multimodal postoperative analgesia will be provided according to institutional protocol
  Interventions: Other: No Regional Block (Control)

INTERVENTIONS:
Procedure: Serratus Plane Block — "Ultrasound-guided serratus anterior plane block performed preoperatively while patients are awake. A total of 30 mL of local anesthetic solution (5 mL saline, 5 mL of 2% lidocaine, 20 mL of 0.25% bupivacaine) will be used. The total volume will be divided equally between both breasts (15 mL per side), with one injection point on each side at the midaxillary line
  Arms: Serratus Plane Block
Procedure: Rhomboid Intercostal Plane Block (RIPB) — Ultrasound-guided rhomboid intercostal plane block (RIPB) performed preoperatively while patients are awake, using a total of 30 mL local anesthetic solution (5 mL normal saline, 5 mL of 2% lidocaine, and 20 mL of 0.25% bupivacaine). The total volume will be divided equally between both breasts (15 mL per side), with one injection point on each side between the rhomboid major muscle and the intercostal muscles at the medial border of the scapula around the 5th intercostal level.
  Arms: Rhomboid Intercostal Plane Block
Other: No Regional Block (Control) — Participants in this group will not receive any regional block. Standard general anesthesia and multimodal postoperative analgesia will be provided according to institutional protocol.
  Arms: Control Group (No Block)

SUMMARY:
This prospective, randomized clinical study aims to compare the analgesic efficacy of serratus plane block (SPB) and rhomboid intercostal plane block (RIPB) for postoperative analgesia in patients undergoing elective bilateral breast reduction surgery under general anesthesia. All patients will receive standardized general anesthesia. Before induction of anesthesia, while patients are awake, Group SPB will receive an ultrasound-guided serratus anterior plane block and Group RIPB will receive an ultrasound-guided rhomboid intercostal plane block. Postoperative analgesia will be maintained with intravenous patient-controlled analgesia (PCA) with opioids. Primary outcomes include postoperative pain scores and opioid consumption at 1, 6, 12, and 24 hours. Secondary outcomes include time to first analgesic demand, patient satisfaction, and block-related complications.

DETAILED DESCRIPTION:
Postoperative pain management in breast reduction surgery is challenging due to wide tissue dissection and thoracic wall involvement. Serratus plane block (SPB) and rhomboid intercostal plane block (RIPB) are regional anesthesia techniques that provide analgesia by blocking the lateral cutaneous branches of the intercostal nerves.

This randomized controlled trial will compare the analgesic efficacy of SPB and RIPB in female patients aged 18-65 undergoing elective bilateral breast reduction surgery under general anesthesia.

Before induction of general anesthesia, while patients are awake, ultrasound-guided SPB or RIPB will be performed according to group allocation. After block performance, general anesthesia will be induced using a standardized protocol. Postoperative pain management will be provided with intravenous patient-controlled analgesia (PCA) with opioids.

Primary outcomes include postoperative pain scores (NRS) and opioid consumption. Secondary outcomes include duration of analgesia, time to first analgesic request, patient satisfaction, and block-related complications. The hypothesis is that both blocks will reduce postoperative pain and opioid consumption, but the duration and quality of analgesia may differ between SPB and RIPB.

ELIGIBILITY:
Inclusion Criteria:

* Female patients aged 18-65 years

American Society of Anesthesiologists (ASA) physical status I-II

Scheduled for elective bilateral breast reduction surgery under general anesthesia

Willing and able to provide written informed consent

Exclusion Criteria:

* Allergy or contraindication to local anesthetics (bupivacaine)

Coagulopathy or anticoagulant medication use

Infection at or near the injection site

History of chronic opioid use or psychiatric/neurological disorders affecting pain perception

Body mass index (BMI) > 35 kg/m²

Refusal to participate in the study

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Only biologically female patients undergoing elective breast reduction surgery will be eligible to participate in this study
Enrollment: 90 (Estimated)
Dates: Start 2025-02-02 (Actual); Primary Completion 2026-02-15 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Postoperative Pain Score at Rest and During Movement at 1, 6, 12, and 24 Hours | 24 hours after surgery
  Pain intensity will be assessed using the Numeric Rating Scale (NRS), a 0-10 point scale where 0 = no pain and 10 = worst imaginable pain. Higher scores indicate worse pain. Pain scores will be recorded at rest and during movement at 1, 6, 12, and 24 hours after surgery. All patients will receive intravenous patient-controlled analgesia (PCA) for postoperative pain management.

CONTACTS AND LOCATIONS:
Overall Officials: Konul karaja, MD, Principal Investigator — Aydın Adnan Menderes University Hospita
Locations (1):
- Aydın Adnan Menderes University Hospital, Department of Anesthesiology and Reanimation, Aydin, Aydın, Turkey (Türkiye)